CLINICAL TRIAL: NCT03034746
Title: Impact of Physical Activity on Successful Aging: Multidisciplinary Analysis of Mechanisms and Outcomes
Brief Title: Impact of Physical Activity on Successful Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, prof. Federico Schena, MD Full Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRIN_2010
Record Dates: First submitted 2017-01-10; First posted 2017-01-27 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer Disease; Cognitive Impairment; Physical Activity
Keywords: alzheimer's disease, physical activity, cognitive training
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Alzheimer's Disease (G1) (Experimental): (G1) physical activity (PA)
  Interventions: Other: Physical activity (PA)
- Alzheimer's Disease (G2) (Experimental): (G2) cognitive treatment (CT)
  Interventions: Other: cognitive treatment (CT)
- Healthy Old Subjects (G1) (No Intervention): Control group old
- Healthy young Subjects (G2) (No Intervention): Control group young

INTERVENTIONS:
Other: Physical activity (PA) — It will perform a program consist of 15 min of warm-up, 60 min of aerobic and resistance training, and 15 min of cool-down.
  Arms: Alzheimer's Disease (G1)
Other: cognitive treatment (CT) — The cognitive stimulation group will received a rehabilitation program with multimodal repetitive stimulation in order to exercise and reinforce the cognitive skills of the participant to slow/prevent the decline. In particular the treatment will be focused on reorient the patient about his/her-self, his/her history and his/her environment, to improve the memory skill by teaching compensatory and restitutive strategies, to help the patient to the discussion about everyday life and in particular to the everyday problems
  Arms: Alzheimer's Disease (G2)

SUMMARY:
Emerging literature suggests that vascular factors might be involved in the pathogenesis of Alzheimer's disease (AD). Other recent studies demonstrate the positive effects of physical activity on cognitive and behavioral disturbances of patients with AD. Therefore, it has been postulated that exercise enchantment in cerebral circulation is the physiological mechanism that link physical exercise and reduction of AD symptoms. Consequently, a program of physical activity could be considered one approach to counteract dementia by improving cerebrovascular health.

However at this moment, it is not clear if the progressive brain vascular dysfunction and hypoperfusion, associated with the β-amyloid deposition, might be reversed or stabilized by an exercise intervention.

The aim of this study is to assess, in patients with AD, the influence of physical exercise, compared to cognitive stimulation, on:

* Cognitive function;
* Independence in daily living and behavioral symptoms;
* Vascular function Finally, to investigate the physiological processes on the basis of the motor parameters' changes, the performances of the patients will be compared with the performances of healthy young and old subjects.

MAIN OBJECTIVE: Investigate, in patients with Mild Cognitive Impairment (MCI) and AD, the effects of a physical activity program, or cognitive stimulation on global cognitive function.

SECONDARY OBJECTIVES: Investigate the effects of the two treatments on:

* cognitive and motor performances,
* independence in activities of daily living,
* behavioral symptoms,
* peripheral vascular function.

DETAILED DESCRIPTION:
STUDY DESIGN:

Randomised controlled, blinded clinical trial.

SUBJECTS:

The study will include 120 patients with definite diagnosis of MCI or AD and 30 young healthy subjects and 30 old healthy subjects referred to the Research Unit associated with the Department.

Patients will be regarded as suitable to participate if they fulfilled the following criteria:

* Mini Mental State Examination (MMSE) ≥ 8;
* Performance Oriented Mobility Assessment ≥ 19 (POMA).

Exclusion criteria will be:

* presence of other concurrent neurological diseases;
* presence of other orthopaedic diseases involving the lower limbs and/or interfering with standing position and/or walking;
* presence of severe auditory and visual deficits not corrected;
* abuse of alcohol or drugs;
* psychiatric disorders,
* severe behavioral disorders;
* hearth and respiratory disease that interfere with the motor activity. The protocol was be approved by the local ethics committee with number 2389. All participants will perform a physiatric examination by a medical doctor of the Department of Neurological and Movement Sciences. Written inform consent will be obtained from all participants before inclusion in the study.

Participants who will meet the inclusion criteria will conduct a clinical and instrumental evaluation at enrollment (T0) and after 6 months ± 15 days after the first visit (T1). The assessment procedures will also be repeated after 3 months (T2) from T1.

ASSESSMENT PROCEDURES

Primary endpoints:

- score obtained in the Mini Mental State Examination.

Secondary endpoints:

- score obtained in a cognitive battery.

For MCI patients will be used:

* Trial Making Test (Reitan,1958),
* Rivermead Behavioral Memory Test (Wilson, 1989),
* Tower of London (Shallice, 1982),
* Dual Task (Della Sala et al., 1997),
* Frontal Assessment Battery (Iavarone A et al., 2004).

For AD patients will be used:

* Attention Matrix (Spinnler et al., 1987),
* Alzheimer's Disease Assessment Scale (Rosen WG et al., 1984),
* Frontal Assessment Battery (Iavarone A et al., 2004).

  - score obtained in a motor skills assessment composed by:
* 6-Minute Walking Test (Ries JD et al., 2009),
* gait analysis by GAITRite® System (Bilney B et al., 2003),
* stabilometric assessments with Stability Line (Nashner LM and Peters JF, 1990),

  * score obtained in the test Instrumental Activity in Daily Living (Lawton MP and Brody EM, 1969),
  * score obtained in the test Neuropsychiatric Inventory (Cummings JL et al., 1994),
  * peripheral vascular function measured by doppler.

To evaluate the effectiveness of motor treatment, compared to a cognitive treatment on motor skills, cognitive skills, behavioral and autonomy in patients with cognitive decline, all patients will be evaluated by motor, cognitive, behavioral and autonomy scales, at baseline, after 6 months (T1), and after others 3 months (T2). A subgroup of 50% of patients will undergo instrumental procedures to investigate the effects of treatments on cerebral blood flow (arterial spin labeling).

TREATMENT PROCEDURES

The participants will be recruited and randomly assigned, according to the degree of cognitive decline, to one of the 3 groups (7-8 subjects):

* Physical Activity group (PA group): It will perform a program consist of 15 min of warm-up, 60 min of aerobic and resistance training, and 15 min of cool-down.
* Cognitive treatment group (CT group): The cognitive stimulation group will received a rehabilitation program with multimodal repetitive stimulation in order to exercise and reinforce the cognitive skills of the participant to slow/prevent the decline. In particular the treatment will be focused on reorient the patient about his/her-self, his/her history and his/her environment, to improve the memory skill by teaching compensatory and restitutive strategies, to help the patient to the discussion about everyday life and in particular to the everyday problems The PA and CT groups will be homogeneous for clinical and demographic data, and participants will undergo 72 treatment group sessions, 60-minute/session, and 3 days/week for 6 consecutively months.

Both types of treatment will be balanced with different degrees of difficulty depending on the state of disease severity .

o The control groups (CG) will not receive any such treatment during the study and they will be evaluated by the same clinical and instrumental assessments.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years;
* Mini Mental State Examination (MMSE) ≥ 8;
* Performance Oriented Mobility Assessment ≥ 19 (POMA).

Exclusion Criteria:

* presence of other concurrent neurological diseases;
* presence of other orthopaedic diseases involving the lower limbs and/or interfering with standing position and/or walking;
* presence of severe auditory and visual deficits not corrected;
* abuse of alcohol or drugs;
* psychiatric disorders,
* severe behavioral disorders;
* hearth and respiratory disease that interfere with the motor activity.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination | 0-6-9 months (change will be assessed)

SECONDARY OUTCOMES:
Trail Making Test | 0-6-9 months (change will be assessed)
  For MCI patients (Reitan,1958)
Rivermead Behavioral Memory Test | 0-6-9 months (change will be assessed)
  For MCI patients (Wilson, 1989)
Tower of London | 0-6-9 months (change will be assessed)
  For MCI patients (Shallice, 1982)
Dual Task | 0-6-9 months (change will be assessed)
  For MCI patients (Della Sala et al., 1997)
Frontal Assessment Battery | 0-6-9 months (change will be assessed)
  (Iavarone A et al., 2004)
Attention Matrix | 0-6-9 months (change will be assessed)
  For AD patients (Spinnler et al., 1987)
Alzheimer's Disease Assessment Scale | 0-6-9 months (change will be assessed)
  For AD patients (Rosen WG et al., 1984)
6-Minute Walking Test | 0-6-9 months (change will be assessed)
  (Ries JD et al., 2009)
gait analysis by GAITRite® System | 0-6-9 months (change will be assessed)
  (Bilney B et al., 2003)
stabilometric assessments with Stability Line | 0-6-9 months (change will be assessed)
  (Nashner LM and Peters JF, 1990),
Instrumental Activity in Daily Living Scale (IADL) | 0-6-9 months (change will be assessed)
Neuropsychiatric Inventory Scale (NPI) | 0-6-9 months (change will be assessed)
cerebral circulation | 0-6-9 months (change will be assessed)
  measured MRI arterial spin labeling
peripheral vascular function | 0-6-9 months (change will be assessed)
  measured by vascular doppler

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, Study Chair — Department of Neurological and Movement Sciences; Federico Schena, Principal Investigator — Department of Neurological and Movement Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Venturelli M, Lanza M, Muti E, Schena F. Positive effects of physical training in activity of daily living-dependent older adults. Exp Aging Res. 2010 Apr;36(2):190-205. doi: 10.1080/03610731003613771. PMID 20209421
- [Result] Venturelli M, Scarsini R, Schena F. Six-month walking program changes cognitive and ADL performance in patients with Alzheimer. Am J Alzheimers Dis Other Demen. 2011 Aug;26(5):381-8. doi: 10.1177/1533317511418956. Epub 2011 Aug 17. PMID 21852281
- [Result] Venturelli M, Magalini A, Scarsini R, Schena F. From Alzheimer's disease retrogenesis: a new care strategy for patients with advanced dementia. Am J Alzheimers Dis Other Demen. 2012 Nov;27(7):483-9. doi: 10.1177/1533317512459794. Epub 2012 Sep 13. PMID 22984089
- [Result] Venturelli M, Scarsini R, Muti E, Salvagno GL, Schena F. Sundowning syndrome and hypothalamic-pituitary-adrenal axis dysregulation in individuals with Alzheimer's disease: is there an association? J Am Geriatr Soc. 2013 Nov;61(11):2055-6. doi: 10.1111/jgs.12491. No abstract available. PMID 24219216
- [Result] Venturelli M, Ce E, Limonta E, Muti E, Scarsini R, Brasioli A, Schena F, Esposito F. Possible Predictors of Involuntary Weight Loss in Patients with Alzheimer's Disease. PLoS One. 2016 Jun 27;11(6):e0157384. doi: 10.1371/journal.pone.0157384. eCollection 2016. PMID 27347878
- [Result] Venturelli M, Sollima A, Ce E, Limonta E, Bisconti AV, Brasioli A, Muti E, Esposito F. Effectiveness of Exercise- and Cognitive-Based Treatments on Salivary Cortisol Levels and Sundowning Syndrome Symptoms in Patients with Alzheimer's Disease. J Alzheimers Dis. 2016 Jul 14;53(4):1631-40. doi: 10.3233/JAD-160392. PMID 27540967
- [Result] Crispoltoni L, Stabile AM, Pistilli A, Venturelli M, Cerulli G, Fonte C, Smania N, Schena F, Rende M. Changes in Plasma beta-NGF and Its Receptors Expression on Peripheral Blood Monocytes During Alzheimer's Disease Progression. J Alzheimers Dis. 2017;55(3):1005-1017. doi: 10.3233/JAD-160625. PMID 27802234
- [Derived] Pedrinolla A, Venturelli M, Tamburin S, Fonte C, Stabile AM, Galazzo IB, Ghinassi B, Venneri MA, Pizzini FB, Muti E, Smania N, Di Baldassarre A, Naro F, Rende M, Schena F. Non-Abeta-Dependent Factors Associated with Global Cognitive and Physical Function in Alzheimer's Disease: A Pilot Multivariate Analysis. J Clin Med. 2019 Feb 9;8(2):224. doi: 10.3390/jcm8020224. PMID 30744116
- [Derived] Pedrinolla A, Venturelli M, Fonte C, Munari D, Benetti MV, Rudi D, Tamburin S, Muti E, Zanolla L, Smania N, Schena F. Exercise Training on Locomotion in Patients with Alzheimer's Disease: A Feasibility Study. J Alzheimers Dis. 2018;61(4):1599-1609. doi: 10.3233/JAD-170625. PMID 29376858